CLINICAL TRIAL: NCT05453812
Title: Meaning of Recovery to Patients Undergoing Lung Cancer Surgery: A Prospective Observational Study
Brief Title: Meaning of Recovery After Lung Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, Clinical Assistant Professor, Seoul National University Hospital
Other Study IDs: Recovery_lung
Record Dates: First submitted 2022-07-03; First posted 2022-07-12 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Recovery; Lung Cancer; Surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to find out the meaning of recovery after lung cancer surgery from a patient's point of view. The results of this study would help improve postoperative recovery in lung cancer patients.

DETAILED DESCRIPTION:
In patients undergoing video-assisted thoracic surgery (VATS) lung resection for lung cancer, the survey on the 'meaning of recovery after surgery' are conducted before surgery, 2 days after surgery, and 30 days after surgery. The questionnaire includes importance score of each question regarding the meaning of recovery after lung cancer surgery.

After 2 days of surgery and 30 days after surgery, the questionnaire about the recovery score and the part where the patients felt difficulties are conducted to investigate what recovery means from a patient's point of view. Length of hospital and ICU stay and postoperative complications are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 80 years undergoing video-assisted thoracic surgery (VATS) lung resection for lung cancer
* Patients who can provide written consent to participate in clinical trials, understand the procedures of this clinical trial, and properly fill out patient-reported questionnaires or respond appropriately to interviews

Exclusion Criteria:

* Patients who did not consent to the trial
* Patients who have difficulty filling out questionnaires or answering interviews about the meaning of recovery
* Patients judged to be inappropriate for this clinical trial based on the opinion of the investigator or investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 19 to 80 years undergoing video-assisted thoracic surgery (VATS) lung resection for lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Importance score of each question regarding the meaning of recovery after lung cancer surgery before surgery | 1 day before surgery
  Importance score of each question regarding the meaning of recovery after lung cancer surgery. The survey includes questions about returning to daily life, resolution of symptoms, overcoming mental strains, regaining independence, and enjoying life. Each question is evaluated on a scale of 1-5, higher number means more importance to the patient.
Importance score of each question regarding the meaning of recovery after lung cancer surgery at postoperative day 2 | postoperative day 2
  Importance score of each question regarding the meaning of recovery after lung cancer surgery. The survey includes questions about returning to daily life, resolution of symptoms, overcoming mental strains, regaining independence, and enjoying life. Each question is evaluated on a scale of 1-5, higher number means more importance to the patient.
Importance score of each question regarding the meaning of recovery after lung cancer surgery at postoperative day 30 | postoperative day 30 (between day 25 and 35)
  Importance score of each question regarding the meaning of recovery after lung cancer surgery. The survey includes questions about returning to daily life, resolution of symptoms, overcoming mental strains, regaining independence, and enjoying life. Each question is evaluated on a scale of 1-5, higher number means more importance to the patient.

SECONDARY OUTCOMES:
Recovery score (0~100 scale) | postoperative day 2, and postoperative day 30 (between day 25 and 35)
  Patient self-assessed recovery score (0-100 scale, higher number means better recovery)
Recovery score evaluated with 15-item Quality of Recovery (QoR-15K) scale | postoperative day 2
  Recovery score evaluated with QoR-15K scale (0-150 scale, higher number means better recovery)
Length of hospital stay (day) | Hospital discharge, an average of 3 days
  Days from the end of surgery to discharge
Length of ICU stay (day) | ICU discharge, an average of 1 day
  Days from the end of surgery to ICU discharge
Postoperative complication | Postoperative day 30
  Postoperative complication related to surgery until postoperative day 30

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea